CLINICAL TRIAL: NCT03465748
Title: Effectiveness of Orthokeratology in Myopia Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Illinois College of Optometry (Other)
Collaborators: Wesley Research Institute (Other)
Responsible Party: Principal Investigator, Jennifer Harthan OD, Chief, Cornea Center for Clinical Excellence, Illinois College of Optometry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15021
Record Dates: First submitted 2018-03-06; First posted 2018-03-14 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental-OrthoK (Experimental): The study will be a randomized control study using a single-masked design to investigate axial elongation and myopic progression in children wearing ortho-k lenses (study group) versus single-vision spectacles or soft contact lenses (control group) for a period of 24 months. A minimum of 40 and a maximum of 60 subjects will be recruited from patients at Illinois Eye Institute. Once eligibility has been determined by an unmasked observer, patients will be randomly assigned to either the orthokeratology group or the single-vision contact lens /spectacle group
  Interventions: Device: OrthoK
- Control (No Intervention): The study will be a randomized control study using a single-masked design to investigate axial elongation and myopic progression in children wearing ortho-k lenses (study group) versus single-vision spectacles (control group) for a period of 24 months. A minimum of 40 and a maximum of 60 subjects will be recruited from patients at Illinois Eye Institute. Once eligibility has been determined by an unmasked observer, patients will be randomly assigned to either the orthokeratology group or the single-vision contact lens /spectacle group

INTERVENTIONS:
Device: OrthoK — orthok (orthokeratology) is the science of changing the curvature or shape of the cornea to change how light is focused on the retina at the back of one's eye. Specially designed molding retainer contact lenses are placed on the eye at night and are removed upon awakening.
  Arms: Experimental-OrthoK

SUMMARY:
The high prevalence of myopia - especially in Asian countries - is well documented, as are the sight-threatening complications of high or degenerative myopia. Retinal detachment, glaucoma, vitreal degeneration and focal retinal changes may occur secondary to the progressive axial elongation of the eye with age. Specialty rigid lenses have long been shown to lessen this progression in the pediatric population; orthokeratology (ortho-k) lenses are worn at night and change the corneal topography to correct low to moderate amounts of myopia. Most of the studies on orthokeratology were conducted on Asian children. To the best of the investigators knowledge, no study has been done on African American (AA) children. The investigators' project seeks to investigate the efficacy of ortho-k in slowing axial elongation and myopic progression in AA children compared to that in other races.

DETAILED DESCRIPTION:
Orthokeratology (ortho-k), when used for partial or full correction of myopia, has been shown to slow myopic progression in children by 36-56% as compared to their spectacle or contact-lens wearing peers.1 This effect is achieved by limiting the axial elongation of the eye,1, 2,3, 4 which is of particular concern in high myopes (>6.00D) and children, where myopic progression has been shown to proceed at a faster rate than average.1 As early intervention is considered beneficial if not essential, Ortho-k as a treatment modality for diminishing myopic progression has, to our knowledge, been studied mostly in Asian children.

The safety and efficacy of ortho-k as a means of decreasing myopic progression was well established by the Children's Overnight Orthokeratology Investigation (COOKI), who evaluated refractive error, visual changes and ocular health over a period of 6 months in myopic children. 7 The Longitudinal Orthokeratology Research in Children (LORIC) study looked at axial elongation in children as old as 12 years, and found that ortho-k decreased axial elongation by approximately 50% compared to be-spectacled controls. 2 They also noted, however, high variability amongst the children that limits the clinician's ability to predict the outcome of the intervention.2 The Corneal Reshaping and Yearly Observation of Myopia (CRAYON) study confirmed that patients fit with ortho-k lenses showed less change in axial length and vitreous chamber depth when compared to subjects wearing soft contact lenses. 3 Other more recent studies by Santodomingo-Rubido et al, 7 Kakita et al4 and Charm et al1 confirm this decrease in axial elongation using IOL Master measurements.

The most commonly accepted theory on how orthokeratology decreases axial elongation relies on the peripheral defocus created on the retina by the corneal changes made by the rigid lens. 9 Hoogerheide et al showed that those at greatest risk for myopic progression were those whose peripheral refraction was hypermetropic10 - that is, they had a hyperopic peripheral 'defocus'. A number of studies have since suggested that treatment approaches to myopia correction should address this peripheral refraction as a means of slowing further axial elongation.9 When looking at subjects treated with ortho k, we see that the lenses do in fact introduce a peripheral myopic defocus while leaving the central refraction more or less emmetropic. 9 With this study, the investigators hope to expand potential application of orthokeratology to a novel population, AA children.

ELIGIBILITY:
Inclusion Criteria:

* myopia progression more than -1.00D in one year
* myopic prescription between -1.00D and -6.00D in at least one eye with refractive astigmatism <1.50D
* Best corrected VA 20/25 or better
* subjects willing to present to clinic for all necessary follow up care
* willing to be randomized to either group

Exclusion Criteria:

* non-compliance with treatment protocol
* contraindications for orthok as per company guidelines
* history of refractive surgery
* current gas permeable contact lens wearers

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Pang, OD, Study Chair — Illinois College of Optometry
Locations (1):
- Illinois Eye Institute, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charm J, Cho P. High myopia-partial reduction ortho-k: a 2-year randomized study. Optom Vis Sci. 2013 Jun;90(6):530-9. doi: 10.1097/OPX.0b013e318293657d. PMID 23645372
- [Background] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Background] Walline JJ, Jones LA, Sinnott LT. Corneal reshaping and myopia progression. Br J Ophthalmol. 2009 Sep;93(9):1181-5. doi: 10.1136/bjo.2008.151365. Epub 2009 May 4. PMID 19416935
- [Background] Kakita T, Hiraoka T, Oshika T. Influence of overnight orthokeratology on axial elongation in childhood myopia. Invest Ophthalmol Vis Sci. 2011 Apr 6;52(5):2170-4. doi: 10.1167/iovs.10-5485. PMID 21212181
- [Background] Loman J, Quinn GE, Kamoun L, Ying GS, Maguire MG, Hudesman D, Stone RA. Darkness and near work: myopia and its progression in third-year law students. Ophthalmology. 2002 May;109(5):1032-8. doi: 10.1016/s0161-6420(02)01012-6. PMID 11986114
- [Background] Kinge B, Midelfart A. Refractive changes among Norwegian university students--a three-year longitudinal study. Acta Ophthalmol Scand. 1999 Jun;77(3):302-5. doi: 10.1034/j.1600-0420.1999.770311.x. PMID 10406150
- [Background] Walline JJ, Rah MJ, Jones LA. The Children's Overnight Orthokeratology Investigation (COOKI) pilot study. Optom Vis Sci. 2004 Jun;81(6):407-13. doi: 10.1097/01.opx.0000135093.77007.18. PMID 15201713
- [Background] Santodomingo-Rubido J, Villa-Collar C, Gilmartin B, Gutierrez-Ortega R. Myopia control with orthokeratology contact lenses in Spain: refractive and biometric changes. Invest Ophthalmol Vis Sci. 2012 Jul 31;53(8):5060-5. doi: 10.1167/iovs.11-8005. PMID 22729437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized control study at the Illinois Eye Institute using a single-masked design to investigate axial elongation and myopic progression in children wearing ortho-k lenses (study group) versus single-vision spectacles or soft contact lenses (control group) for a period of twenty-four months (May 2017 to January 2021) There was a delay in the recruitment and some subjects lost to follow up due to COVID.
Period: Overall Study
Arm/Group | Experimental-OrthoK | Control
Started | 27 | 18
Completed | 15 | 7
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Population: Due to COVID, there were some limitations in recruiting for the study and finishing the enrollment.
Groups:
- Experimental-OrthoK: The study will be a randomized control study using a single-masked design to investigate axial elongation and myopic progression in children wearing ortho-k lenses (study group) versus single-vision spectacles or soft contact lenses (control group) for a period of 24 months. Once eligibility has been determined by an unmasked observer, patients will be randomly assigned to either the orthokeratology group or the single-vision contact lens /spectacle group
  OrthoK: orthok (orthokeratology) is the science of changing the curvature or shape of the cornea to change how light is focused on the retina at the back of one's eye. Specially designed molding retainer contact lenses are placed on the eye at night and are removed upon awakening.
- Control: The study will be a randomized control study using a single-masked design to investigate axial elongation and myopic progression in children wearing ortho-k lenses (study group) versus single-vision spectacles (control group) for a period of 24 months. Once eligibility has been determined by an unmasked observer, patients will be randomly assigned to either the orthokeratology group or the single-vision contact lens /spectacle group.
- Total: Total of all reporting groups
Arm/Group | Experimental-OrthoK | Control | Total
Number analyzed (Participants) | 27 | 18 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 18 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 22 | 17 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 9 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 3 | 1 | 4
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 18 | 45
spherical equivalent refractive error [Mean (Full Range); unit: Diopters] | 2.69 [0.50 to 6.00] | 3.50 [1.50 to 6.00] | 3.18 [0.50 to 6.00]

OUTCOME MEASURES:

1. Primary Outcome: Axial Length
Description: Axial Length was measured at baseline and again at the 2 year mark. Units are given in mm. The average of axial length at the 2 year period is provided.
Time Frame: 2 years
Population: Axial length was measured in mm, many subjects withdrew from the study due to patient/parent scheduling
Measure: Mean (Full Range); unit: mm
Arm/Group | Experimental-OrthoK | Control
Number analyzed (Participants) | 15 | 7
mm | 25.32 [25.07 to 26.23] | 26.08 [25.59 to 26.74]

ADVERSE EVENTS:
Time Frame: At each examination over the course of the 24 month study, subjects were asked about any adverse events.
Description: If any adverse events were identified, subjects were asked to notify the principal investigator.
Arm/Group | Experimental-OrthoK | Control
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/14
Other Adverse Events (participants affected / at risk) | 1/27 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental-OrthoK (N=27) | Control (N=14)
Corneal Binding (Eye disorders) | 1 (1) | 0 (0) — One patient in the treatment arm had corneal binding occur in which the contact lens caused corneal staining and irritation. The patient immediately discontinued lens wear and was treated successfully.

LIMITATIONS AND CAVEATS:
Many subjects withdrew from the study due to scheduling conflicts. There was also a pause towards the end of the study follow up due to COVID. Some subjects withdrew from the study due to not being able to tolerate the lenses. Some subjects lost many lenses and had to re-order repeatedly throughout the study, limiting their success in completing the study. Remote learning during COVID may have impacted myopia progression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT03465748/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT03465748/ICF_001.pdf